CLINICAL TRIAL: NCT06542718
Title: Studying the Heterogeneity of Gestational Diabetes Mellitus: Cardio-Metabolic Alteration and Treatment Response in a Multi-Ethnic Population in Singapore (GDM-CARE)
Brief Title: Studying Phenotypes of Gestational Diabetes Mellitus in an Asian Pregnant Cohort
Acronym: GDM-CARE
Status: Recruiting | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Lingjun Li, Assistant Director, Public Affairs, Global Centre for Asian Women's Health, Assistant Professor, Department of O&G, Yong Loo Lin School of Medicine, National University of Singapore, National University Health System, Singapore
Other Study IDs: 2021/01076
Record Dates: First submitted 2024-07-27; First posted 2024-08-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes; Pregnancy Related; Pregnancy Complications; Birth Weight; Insulin Resistance, Diabetes; Intergenerational Relations
Keywords: Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Birth Weight; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and fecal samples will be collected across gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gestational diabetes mellitus (GDM) is a transient hyperglycemic condition identified during pregnancy in women without a history of chronic diabetes. Evidence indicates that GDM can lead to various adverse health outcomes, including preterm birth, progression to pre-diabetes, and type 2 diabetes after delivery in mothers. Notably, GDM is becoming increasingly prevalent among Asian pregnant women due to rising rates of overweight and obesity, as well as genetic susceptibility. Despite growing recognition of GDM, its treatment efficiency and efficacy remain poor, primarily due to its heterogeneity, which is underpinned by various pathophysiological mechanisms.

Therefore, a better understanding of GDM heterogeneity can aid clinicians in providing more targeted treatment and follow-up strategies for GDM mothers. This study aims to define GDM phenotypes based on in vivo cardio-metabolic profiles and treatment response during pregnancy, utilizing advanced technologies such as continuous glucose profiling and untargeted metabolite profiling. In this proposed 3-year pregnancy cohort study, the investigators will recruit 800 overweight or obese Asian pregnant women in early pregnancy, without a history of diabetes, and follow them through to delivery. The goal of the study is to develop systematic antenatal and postnatal screening, treatment, and intervention guidelines for mothers with GDM.

DETAILED DESCRIPTION:
The transient hyperglycemia first identified during pregnancy is known as gestational diabetes mellitus (GDM). GDM increases the risks of adverse pregnancy and neonatal outcomes, such as pre-eclampsia and macrosomia. Due to the widespread prevalence of overweight, obesity, and genetic susceptibility, GDM is more common among Asian pregnant women-occurring 2- to 3-fold more frequently compared to European pregnant women, with rates ranging from 15% to 30% in individuals of Chinese and Indian descent.

Emerging evidence suggests that variations in insulin sensitivity, fat deposition, and β-cell activity may contribute to the heterogeneous phenotypes of GDM, leading to different pregnancy outcomes and maternal diabetic progression. However, current clinical treatment and follow-up strategies for GDM typically adopt a "one-size-fits-all" approach, ignoring the underlying pathophysiological variations among patients. As a result, the efficiency and efficacy of the current clinical approach during pregnancy and postpartum are suboptimal.

In this study, the investigators aim to define the heterogeneity of GDM in terms of in vivo cardio-metabolic profiling and treatment response during pregnancy, using advanced technologies such as continuous glucose profiling and untargeted metabolite profiling. The investigators hypothesize that a better clinical and molecular understanding of GDM phenotypes will enable tailored, effective treatment strategies for individuals and aid in predicting and preventing postnatal abnormal glucose metabolism.

This proposed 3-year longitudinal study will involve a cohort of 800 overweight (23-24.9 kg/m²) or obese (≥25 kg/m²) singleton pregnant women, recruited no later than 12 weeks of gestation. These women, who are of Chinese, Malay, and Indian ethnicities, will be recruited from the National University Hospital (NUH) in Singapore and will not have a history of diabetes. All participants will be screened for GDM at 24-28 weeks of gestation and followed until delivery.

The primary outcome will be the identification of GDM phenotype-specific continuous glycemic profiles and alterations in cardio-metabolic biomarkers. The secondary outcome will focus on the treatment responses specific to different GDM phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of ≤ 13 weeks 6 days
* Overweight and obese subjects with BMI of 23kg/m² - 24.9kg/m² and ≥ 25.0kg/m², respectively
* Aged 21-45 years with singleton pregnancy
* Plan to be followed up during the whole pregnancy and deliver at NUH
* Chinese, Malay or Indian ethnicity for pregnant subject
* Can complete questionnaires in English language
* Willing to wear continuous glucose monitoring device at least for 7 days at each required clinic visit

Exclusion Criteria:

* Participants who are not Singapore citizens or Singapore Permanent Residents, not intending to eventually deliver in Singapore National University Hospital and to reside in Singapore for the next 2 years
* Have serious skin conditions (eg. eczema) that precludes wearing the sensor for 14 days
* With history of Type 1 diabetes or Type 2 diabetes
* With chronic preexisting life-threatening conditions including pancreatic cancer, end-stage kidney dysfunction, and psychosis
* Unable to read or speak English

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant subjects are recruited in the National University Hospital in Singapore.
Study Population: This is a prospective longitudinal study conducted at the Singapore National University Hospital (NUH) Obstetrics and Gynecology outpatient clinic. A cohort of 800 pregnant women will be recruited at NUH over a period of 18 months. The study involves 800 overweight (23-24.9 kg/m²) or obese (≥25 kg/m²) singleton pregnant women-without a history of diabetes and comprising Chinese, Malay, and Indian ethnicities-during their first trimester at the National University Hospital (NUH) in Singapore. All participants will be recruited no later than 12 weeks of gestation and screened for GDM between 24 and 28 weeks of gestation. The investigators will then follow up with the women diagnosed with GDM (approximately 200) from 32-34 weeks of gestation until delivery.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
IADPSG (International Association of Diabetes and Pregnancy Study Groups)-defined Gestational Diabetes Mellitus (GDM) | 3 years
  Oral Glucose Tolerance Test (OGTT) will be performed during universal screening at 24-28 weeks of gestational age. 0, 1 hour and 2 hour glucose readings will be measured after 8-10 hours of overnight fasting, after a 75 grams glucose drink. Cutoffs are according to The International Association of Diabetes and Pregnancy Study Groups (IADPSG) guidelines.

SECONDARY OUTCOMES:
Rates of Diet or Insulin-treated gestational diabetes mellitus based on phenotypes | 3 years
  The rates of treatment-specific gestational diabetes phenotypes will be calculated.

OTHER OUTCOMES:
Rate of large-for-gestational age (LGA) babies based on GDM phenotypes | 3 year
  The numbers and rates of LGA babies according to different GDM phenotypes will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynaecology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared based on write-in proposal to the PI.

REFERENCES:
- [Background] McIntyre HD, Catalano P, Zhang C, Desoye G, Mathiesen ER, Damm P. Gestational diabetes mellitus. Nat Rev Dis Primers. 2019 Jul 11;5(1):47. doi: 10.1038/s41572-019-0098-8. PMID 31296866
- [Background] Chong YS, Cai S, Lin H, Soh SE, Lee YS, Leow MK, Chan YH, Chen L, Holbrook JD, Tan KH, Rajadurai VS, Yeo GS, Kramer MS, Saw SM, Gluckman PD, Godfrey KM, Kwek K; GUSTO study group. Ethnic differences translate to inadequacy of high-risk screening for gestational diabetes mellitus in an Asian population: a cohort study. BMC Pregnancy Childbirth. 2014 Oct 2;14:345. doi: 10.1186/1471-2393-14-345. PMID 25273851
- [Background] Yu Q, Aris IM, Tan KH, Li LJ. Application and Utility of Continuous Glucose Monitoring in Pregnancy: A Systematic Review. Front Endocrinol (Lausanne). 2019 Oct 11;10:697. doi: 10.3389/fendo.2019.00697. eCollection 2019. PMID 31681170
- [Background] Powe CE, Hivert MF, Udler MS. Defining Heterogeneity Among Women With Gestational Diabetes Mellitus. Diabetes. 2020 Oct;69(10):2064-2074. doi: 10.2337/dbi20-0004. Epub 2020 Aug 25. PMID 32843565

DOCUMENTS (1):
  • Study Protocol (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT06542718/Prot_000.pdf